CLINICAL TRIAL: NCT04676022
Title: A Randomized Controlled Study to Evaluate the Safety and Effectiveness of Boston Scientific Spinal Cord Stimulation (SCS) Systems in the Treatment of Chronic Low Back and/or Leg Pain With No Prior Surgeries
Brief Title: SCS as an Option for Chronic Low Back and/or Leg Pain Instead of Surgery
Acronym: SOLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4077
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
Keywords: Spinal Cord Stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Spinal Cord Stimulation (Experimental): To receive Spinal Cord Stimulation programming
  Interventions: Device: WaveWriter
- Conventional Medical Management (Other): To receive conventional medical management
  Interventions: Other: Conventional Medical Managament

INTERVENTIONS:
Device: WaveWriter — To receive Spinal Cord Stimulation programming
  Arms: Spinal Cord Stimulation
Other: Conventional Medical Managament — To receive conventional medical management
  Arms: Conventional Medical Management

SUMMARY:
To evaluate the safety and effectiveness of Spinal Cord Stimulation (SCS) with multiple modalities compared to Conventional Medical Management (CMM) in patients with chronic low back and/or leg pain who have not undergone spinal surgery when using the Boston Scientific WaveWriter SCS Systems.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic low back pain, with or without leg pain, for at least 6 months
* Received at least 90 days of documented pain management care to address the primary pain complaint, prior to Screening (e.g. medication, physical therapy)
* If female of childbearing potential: not pregnant, as evidenced by a negative pregnancy test at Screening
* Subject signed a valid, IRB-approved informed consent form (ICF) provided in English

Key Exclusion Criteria:

* Primary pain complaint of vascular origin (e.g. peripheral vascular disease)
* Require implantation of lead(s) in the cervical epidural space
* Significant cognitive impairment at Screening that, in the opinion of the Investigator, would reasonably be expected to impair the study candidate's ability to assess pain intensity
* Previous failed spinal cord stimulation trial or is already implanted with an active implantable device(s) (e.g. pacemaker, drug pump, implantable pulse generator)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2025-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Corporation
Locations (23):
- United States (23):
  - Vitamed Research, Palm Desert, California
  - Summit Pain Alliance, Santa Rosa, California
  - Denver Back Pain Specialists, Greenwood Village, Colorado
  - South Lake Pain Institute, Inc, Clermont, Florida
  - University of Chicago Hospital, Chicago, Illinois
  - Goodman Campbell Brain and Spine, Carmel, Indiana
  - Crimson Pain Management, Overland Park, Kansas
  - MedPharmics, LLC, Metairie, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Willis-Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - Forest Health Medical Center, Ypsilanti, Michigan
  - Saint Louis Pain Consultants, Chesterfield, Missouri
  - Weill Cornell Medical University, New York, New York
  - Carolinas Research Institute, PLLC, Huntersville, North Carolina
  - Novant Health-Hawthorne, Winston-Salem, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - The Toledo Clinic, Toledo, Ohio
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - Delaware Valley Pain and Spine Institute, Trevose, Pennsylvania
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - Institute of Precision Pain Medicine, Corpus Christi, Texas
  - Precision Spine Care, Tyler, Texas
  - University of Utah Orthopaedic Center, Salt Lake City, Utah

REFERENCES:
- [Derived] North J, Calodney A, Trainor D, McCormick ZL, Paez J, Loudermilk E, Christopher A, Noles J, Phillips G, Jolly S, Yang MI, Guirguis M, Kloster D, Pak DJ, Peacock J, Engle M, Shah B, Wilson D, Anitescu M, Atallah J, Chatas J, Leier T, Rosen S, Goldberg E. Spinal cord stimulation plus conventional medical management versus conventional medical management alone for severe, non-surgical, refractory back pain: a randomized clinical trial followed by crossover. Reg Anesth Pain Med. 2025 Oct 5:rapm-2024-106335. doi: 10.1136/rapm-2024-106335. Online ahead of print. PMID 41047246
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 241 subjects provided informed consent.
Pre-assignment Details: After subjects were consented and enrolled, they were evaluated per study eligibility criteria. Only those who met criteria proceeded to randomization.
Groups:
- Spinal Cord Stimulation: Randomized to receive Spinal Cord Stimulation programming
  WaveWriter: To receive Spinal Cord Stimulation programming
- Conventional Medical Management: Randomized to receive conventional medical management
  Conventional Medical Managament: To receive conventional medical management
- Non-randomized Subjects: Consented subjects who were not randomized in the study.
Period: Overall Study
Arm/Group | Spinal Cord Stimulation | Conventional Medical Management | Non-randomized Subjects
Started | 79 | 68 | 94
Completed | 57 | 64 | 0
Not Completed | 22 | 4 | 94
Not completed — Screen Failure/ | 1 | 1 | 85
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 6
Not completed — Will not move forward with permanent implant | 6 | 0 | 0
Not completed — Various reasons (moved, no longer meets criteria, visit not done etc.) | 7 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized subjects
Groups:
- Randomized to Spinal Cord Stimulation (SCS) Treatment Activated: Baseline demographics and clinical characteristics for subjects in the SCS arm
- Randomized to Conventional Medical Management (CMM) Treatment Activated: Baseline demographics and clinical characteristics for subjects in the CMM arm
- Total: Total of all reporting groups
Arm/Group | Randomized to Spinal Cord Stimulation (SCS) Treatment Activated | Randomized to Conventional Medical Management (CMM) Treatment Activated | Total
Number analyzed (Participants) | 79 | 68 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (12.10) | 61.0 (11.9) | 59.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 43 | 98
  Male | 24 | 25 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity : American Indian or Alaska native | 0 | 1 | 1
  Race and Ethnicity : Black, of African heritage | 6 | 3 | 9
  Race and Ethnicity : Caucasian | 72 | 62 | 134
  Race and Ethnicity : Not disclosed | 1 | 0 | 1
  Race and Ethnicity : Hispanic or Latino | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 79 | 68 | 147
Duration of Low Back Pain [Mean (Standard Deviation); unit: years] | 11.5 (10.4) | 12.9 (11.5) | 12.2 (10.9)
Average low back pain (VRS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity is expressed on a 0 - 10 verbal rating scale (VRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine".
  units on a scale | 7.5 (1.0) | 7.6 (0.9) | 7.6 (0.9)
Average overall pain (VRS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity is expressed on a 0 - 10 verbal rating scale (VRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine".
  units on a scale | 7.5 (0.9) | 7.5 (1.0) | 7.5 (0.9)
Oswestry Disability Index (ODI) Summary Score [Mean (Standard Deviation); unit: units on a scale] — Change in Disability (Oswestry Disability Index). The Oswestry Disability Index (ODI) is a validated questionnaire of pain-related disability with total score on a scale of 0 (no disability) to 100 (complete disability). Categories for ODI total score are 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The published minimally clinically important difference for change in ODI is 10 points.
  units on a scale | 54.4 (8.5) | 54.4 (9.4) | 54.4 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate
Description: Proportion of subjects with 50% or greater reduction in overall pain relief
Time Frame: 3 months post-activation
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Cord Stimulation | Conventional Medical Management
Number analyzed (Participants) | 57 | 62
Participants | 51 | 5

2. Secondary Outcome: Change in Disability (Oswestry Disability Index)
Description: Change in Disability (Oswestry Disability Index). The Oswestry Disability Index (ODI) is a validated questionnaire of pain-related disability with total score on a scale of 0 (no disability) to 100 (complete disability). Categories for ODI total score are 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The published minimally clinically important difference for change in ODI is 10 points.
Time Frame: 3-Months post activation
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spinal Cord Stimulation | Conventional Medical Management
Number analyzed (Participants) | 57 | 64
score on a scale | -27.5 (15.9) | -7.2 (9.9)

ADVERSE EVENTS:
Time Frame: Randomized subjects through 3-Months post-Activation, an average of 6 months.
Groups:
- Randomized to SCS: Subjects Randomized to SCS Arm through 3 Months post-Activation.
- Randomized to CMM: Subjects Randomized to CMM Arm through 3 Months post-Activation.
Arm/Group | Randomized to SCS | Randomized to CMM
All-Cause Mortality (participants affected / at risk) | 0/79 | 1/68
Serious Adverse Events (participants affected / at risk) | 8/79 | 1/68
Other Adverse Events (participants affected / at risk) | 9/79 | 4/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to SCS (N=79) | Randomized to CMM (N=68)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Alcohol Use Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to SCS (N=79) | Randomized to CMM (N=68)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT04676022/Prot_SAP_000.pdf